CLINICAL TRIAL: NCT03259191
Title: Department of Gastroenterology, Zhongda Hospital
Brief Title: Anti-reflux Mucosectomy (ARMS) is a Useful Therapy for Refractory Gastroesophageal Reflux Disease (RGERD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruihua Shi (Other)
Responsible Party: Sponsor-Investigator, Ruihua Shi, MD, PhD, Postdoctoral Mentor, Chief Physician, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GI of Zhongda
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Refractory Gastroesophageal Reflux Disease
Keywords: Anti-reflux mucosectomy,refractory gastroesophageal reflux disease,safety,efficacy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- completely circumferential ARMS (Other)
  Interventions: Procedure: anti-reflux mucosectomy
- semi-circumferential ARMS (Other)
  Interventions: Procedure: anti-reflux mucosectomy

INTERVENTIONS:
Procedure: anti-reflux mucosectomy — Anti-reflux mucosectomy (ARMS) may be a new therapy for refractory gastroesophageal reflux disease (RGERD). The aim of the present study is to explore the safety and efficacy of ARMS.

SUMMARY:
Anti-reflux mucosectomy (ARMS) may be a new therapy for refractory gastroesophageal reflux disease (RGERD). The aim of the present study is to explore the safety and efficacy of ARMS.

ELIGIBILITY:
Inclusion Criteria:

1. Full sufficiency in literacy
2. Be off proton pump inhibitor, antacids and prokinetics ≥ 2 weeks
3. Refractory gastroesophageal reflux disease

Exclusion Criteria:

1. Severe heart, lung, and cerebrovascular disease
2. Severe hematopoietic system disease
3. Abnormal blood coagulation function
4. Oropharyngeal abnormalities
5. Severe spine malformation
6. In pregnancy and lactation at present, or plan to become pregnant within 2 years
7. Severe inflammation or huge ulcers in stomach
8. Mental and psychological disorde

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-11-20 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms | 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Improvement of all the symptoms related with RGERD.

SECONDARY OUTCOMES:
Complications of ARMS | 1 month, 3 months, 6 months, 12 months, 18 months, 24 months, 30 months, 36 months
  Complications of ARMS,such as esophageal stenosis and dysphagia.

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Wang, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No